CLINICAL TRIAL: NCT01949090
Title: An Observer-blind Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Influenza Vaccine(s) GSK2789869A Administered in Adults 65 Years of Age and Older
Brief Title: Immunogenicity and Safety Study of Different Formulations of GlaxoSmithKline (GSK) Biologicals H7N1 Influenza Vaccine Administered to Adults 65 Years of Age and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200613
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Influenza
Keywords: H7N1; AS03 adjuvant; Safety; Immunogenicity; Influenza; Adults; Elderly adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- GSK2789869A F1 Group (Experimental): Healthy male and female adults, 65 years of age and older, who received two doses of GSK2789869A H7N1 vaccine Formulation 1 (F1), administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- GSK2789869A F2 Group (Experimental): Healthy male and female adults, 65 years of age and older, who received two doses of GSK2789869A H7N1 vaccine Formulation 2 (F2), administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- GSK2789869A F3 Group (Experimental): Healthy male and female adults, 65 years of age and older, who received two doses of GSK2789869A H7N1 vaccine Formulation 3 (F3), administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- GSK2789869A F4 Group (Experimental): Healthy male and female adults, 65 years of age and older, who received two doses of GSK2789869A H7N1 vaccine Formulation 4 (F4), administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- Placebo Group (Placebo Comparator): Healthy male and female adults, 65 years of age and older, who received two doses of Placebo, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Investigational H7N1 vaccine GSK2789869A — Two doses of GSK2789869A H7N1 vaccine administered intramuscularly to the deltoid region at Day 0 and Day 21.
  Arms: GSK2789869A F1 Group; GSK2789869A F2 Group; GSK2789869A F3 Group; GSK2789869A F4 Group
Biological: Placebo — Two doses of placebo administered intramuscularly to the deltoid region at Day 0 and Day 21.
  Arms: Placebo Group

SUMMARY:
The purpose of this placebo controlled study is to evaluate the safety and immunogenicity of different formulations of GSK Biologicals H7N1 influenza vaccine in subjects 65 years of age and older. The study will evaluate safety related events and antibody immune responses to different formulations of study vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults who are 65 years of age and older at the time of first study vaccination.
* Written informed consent obtained from the subject.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Stable health status, as established by medical history and physical exam, and defined by absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within 1 month prior to enrollment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.

Exclusion Criteria:

* Presence or evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence or evidence of substance abuse.
* Diagnosed with cancer, or treatment for cancer within three years.

  * Persons with a history of cancer who are disease-free without treatment for three years or more are eligible.
  * Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and are eligible, but other histologic types of skin cancer are exclusionary.
  * Women who are disease-free three years or more after treatment for breast cancer and receiving long-term prophylaxis are eligible.
* Diagnosed with excessive daytime sleepiness (unintended sleep episodes during the day present almost daily for at least one month), or narcolepsy; or history of narcolepsy in subject's parent, sibling or child.
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 30 days prior to the first dose of study vaccine/placebo, or any other cytotoxic, immunosuppressive or immune-modifying drugs within 6 months of first study vaccine/placebo dose. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or Guillain Barré Syndrome within 42 days of receipt of prior seasonal or pandemic influenza vaccine.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first dose of study vaccine/placebo.
* Planned administration of any vaccine other than the study vaccine/placebo before blood sampling at the Day 42 visit.
* Previous administration of any H7 vaccine or physician-confirmed H7 disease.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period.
* Receipt of any immunoglobulins and/or any blood products within 90 days before the first dose of study vaccine/placebo, or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine including a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 363 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2013-12-04 (Actual); Study Completion 2014-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (5):
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
- Canada (3):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario

REFERENCES:
- [Derived] Madan A, Ferguson M, Rheault P, Seiden D, Toma A, Friel D, Soni J, Li P, Innis BL, Schuind A. Immunogenicity and safety of an AS03-adjuvanted H7N1 vaccine in adults 65years of age and older: A phase II, observer-blind, randomized, controlled trial. Vaccine. 2017 Apr 4;35(15):1865-1872. doi: 10.1016/j.vaccine.2017.02.057. Epub 2017 Mar 13. PMID 28302407

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 363 subjects enrolled in the study, 3 subjects did not receive any vaccination.
Period: Overall Study
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Started | 60 | 60 | 60 | 60 | 120
Completed | 56 | 58 | 58 | 59 | 116
Not Completed | 4 | 2 | 2 | 1 | 4
Not completed — Serious Adverse Event | 0 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1
Not completed — Protocol non-compliance | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group | Total
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.9 (6.0) | 73.9 (6.3) | 73.6 (6.5) | 73.4 (5.3) | 73.0 (5.2) | 73.30 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 30 | 36 | 76 | 214
  Male | 25 | 23 | 30 | 24 | 44 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic Ancestry: African Heritage/African American | 4 | 0 | 5 | 3 | 2 | 14
  Geographic Ancestry: Asian - East Asian Heritage | 0 | 0 | 2 | 0 | 1 | 3
  Geographic Ancestry: Asian - South East Asian Heritage | 0 | 1 | 0 | 0 | 0 | 1
  Geographic Ancestry: White - Arabic/North African Heritage | 0 | 0 | 0 | 0 | 1 | 1
  Geographic Ancestry: White - Caucasian/European Heritage | 56 | 59 | 52 | 57 | 116 | 340
  Geographic Ancestry: Other | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted (SCR) Subjects for Hemagglutination Inhibition (HI) Antibodies Against the Flu A/Mallard/NL/12/2000 (H7N1) Virus Strain
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 10 post-vaccination], antibody titer greater than or equal to (≥) 40 after vaccination; For initially seropositive subjects (antibody titer ≥ 10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/mallard/Netherlands/12/2000 NIBRG-63 (H7N1) (Flu A/mallard/NL/12/2000 H7N1).
Time Frame: At Day 42
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects for whom data concerning immunogenicity outcome measure were available. This primary outcome measure was centered on the groups that received GSK2789869A vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Group: Healthy male and female adults, 65 years of age and older, who received two doses of Placebo, administered intramuscularly in the deltoid region of thee non-dominant arm at Day 0 and of the dominant arm at Day 21.
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 56 | 55 | 53 | 112
Participants | 39 | 45 | 42 | 46 | 0

2. Primary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against the Flu A/Mallard/NL/12/2000 (H7N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection.
Time Frame: At Day 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom data concerning immunogenicity outcome measure were available. This primary outcome measure was centered on the groups that received GSK2789869A vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 56 | 55 | 53 | 112
Participants | 39 | 49 | 43 | 47 | 1

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/Mallard/NL/12/2000 (H7N1) Virus Strain
Description: GMFR, also known as seroconversion factor (SCR) or mean geometric increase (MGI), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer for the vaccine virus.
Time Frame: At Day 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom data concerning immunogenicity outcome measure were available. This primary outcome was centered on the groups that received GSK2789869A vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 56 | 55 | 53 | 112
Fold increase | 11.0 [7.3 to 16.5] | 18.9 [14.0 to 25.4] | 16.0 [10.8 to 23.7] | 18.2 [12.6 to 26.3] | 1.0 [1.0 to 1.1]

4. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest; prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants
  Any Pain, Dose 1 | 27 | 34 | 16 | 29 | 7
  Grade 3 Pain, Dose 1 | 0 | 1 | 0 | 1 | 0
  Any Redness, Dose 1 | 0 | 3 | 1 | 4 | 1
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 1 | 1 | 3 | 2 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 59 | 60 | 58 | 57 | 118
  Any Pain, Dose 2 | 27 | 24 | 17 | 25 | 3
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 59 | 60 | 58 | 57 | 118
  Grade 3 Pain, Dose 2 | 0 | 0 | 2 | 0 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 59 | 60 | 58 | 57 | 118
  Any Redness, Dose 2 | 1 | 1 | 1 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 59 | 60 | 58 | 57 | 118
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 59 | 60 | 58 | 57 | 118
  Any Swelling, Dose 2 | 1 | 2 | 2 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 59 | 60 | 58 | 57 | 118
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 38 | 39 | 25 | 38 | 8
  Grade 3 Pain, Across doses | 0 | 1 | 2 | 1 | 1
  Any Redness, Across doses | 1 | 4 | 1 | 4 | 1
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across doses | 2 | 2 | 4 | 2 | 0
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (symptoms included nausea, vomiting, diarrhoea and/or abdominal pain), headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = temperature > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants
  Any Fatigue, Dose 1 | 7 | 14 | 10 | 8 | 22
  Grade 3 Fatigue, Dose 1 | 1 | 2 | 0 | 0 | 2
  Related Fatigue, Dose 1 | 5 | 8 | 7 | 4 | 13
  Any Fever, Dose 1 | 1 | 1 | 0 | 0 | 0
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 1 | 1 | 0 | 0 | 0
  Any Gastrointestinal, Dose 1 | 5 | 10 | 5 | 6 | 12
  Grade 3 Gastrointestinal, Dose 1 | 1 | 1 | 1 | 0 | 0
  Related Gastrointestinal, Dose 1 | 3 | 4 | 4 | 4 | 7
  Any Headache, Dose 1 | 9 | 13 | 9 | 9 | 19
  Grade 3 Headache, Dose 1 | 1 | 0 | 1 | 0 | 1
  Related Headache, Dose 1 | 7 | 6 | 6 | 4 | 10
  Any Joint pain, Dose 1 | 9 | 3 | 5 | 6 | 14
  Grade 3 Joint pain, Dose 1 | 0 | 0 | 1 | 0 | 1
  Related Joint pain, Dose 1 | 6 | 1 | 3 | 3 | 10
  Any Muscle aches, Dose 1 | 10 | 13 | 5 | 11 | 17
  Grade 3 Muscle aches, Dose 1 | 0 | 1 | 1 | 0 | 1
  Related Muscle aches, Dose 1 | 9 | 11 | 3 | 8 | 12
  Any Shivering, Dose 1 | 3 | 1 | 3 | 1 | 5
  Grade 3 Shivering, Dose 1 | 0 | 0 | 0 | 0 | 1
  Related Shivering, Dose 1 | 3 | 0 | 1 | 0 | 3
  Any Sweating, Dose 1 | 1 | 2 | 3 | 3 | 7
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 0 | 2
  Related Sweating, Dose 1 | 1 | 2 | 0 | 1 | 5
  Any Fatigue, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Fatigue, Dose 2 | 7 | 11 | 7 | 6 | 12
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Fatigue, Dose 2 | 0 | 1 | 1 | 0 | 1
  Related Fatigue, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Fatigue, Dose 2 | 6 | 7 | 5 | 5 | 6
  Any Fever, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Fever, Dose 2 | 0 | 0 | 1 | 0 | 1
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 0 | 1
  Related Fever, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Fever, Dose 2 | 0 | 0 | 1 | 0 | 0
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Gastrointestinal, Dose 2 | 7 | 3 | 6 | 3 | 6
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0 | 2 | 1 | 0
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Gastrointestinal, Dose 2 | 3 | 2 | 3 | 1 | 2
  Any Headache, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Headache, Dose 2 | 8 | 10 | 9 | 6 | 9
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Headache, Dose 2 | 0 | 2 | 1 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Headache, Dose 2 | 6 | 4 | 8 | 5 | 5
  Any Joint pain, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Joint pain, Dose 2 | 4 | 10 | 5 | 5 | 10
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Joint pain, Dose 2 | 0 | 1 | 1 | 0 | 1
  Related Joint pain, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Joint pain, Dose 2 | 3 | 5 | 4 | 4 | 6
  Any Muscle aches, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Muscle aches, Dose 2 | 10 | 12 | 8 | 11 | 11
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Muscle aches, Dose 2 | 0 | 1 | 1 | 0 | 1
  Related Muscle aches, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Muscle aches, Dose 2 | 10 | 9 | 7 | 9 | 8
  Any Shivering, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Shivering, Dose 2 | 3 | 5 | 1 | 2 | 3
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Shivering, Dose 2 | 0 | 1 | 0 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Shivering, Dose 2 | 3 | 2 | 1 | 0 | 2
  Any Sweating, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Any Sweating, Dose 2 | 2 | 4 | 4 | 2 | 1
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Grade 3 Sweating, Dose 2 | 0 | 0 | 1 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 58 | 60 | 58 | 57 | 118
  Related Sweating, Dose 2 | 2 | 3 | 3 | 1 | 1
  Any Fatigue, Across doses | 11 | 19 | 13 | 11 | 28
  Grade 3 Fatigue, Across doses | 1 | 3 | 1 | 0 | 3
  Related Fatigue, Across doses | 8 | 13 | 10 | 8 | 17
  Any Fever, Across doses | 1 | 1 | 1 | 0 | 1
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 1
  Related Fever, Across doses | 1 | 1 | 1 | 0 | 0
  Any Gastrointestinal, Across doses | 11 | 11 | 8 | 9 | 16
  Grade 3 Gastrointestinal, Across doses | 1 | 1 | 2 | 1 | 0
  Related Gastrointestinal, Across doses | 5 | 5 | 5 | 5 | 9
  Any Headache, Across doses | 13 | 17 | 13 | 11 | 24
  Grade 3 Headache, Across doses | 1 | 2 | 1 | 0 | 1
  Related Headache, Across doses | 9 | 9 | 10 | 8 | 13
  Any Joint pain, Across doses | 12 | 12 | 8 | 8 | 17
  Grade 3 Joint pain, Across doses | 0 | 1 | 1 | 0 | 2
  Related Joint pain, Across doses | 8 | 6 | 7 | 5 | 12
  Any Muscle aches, Across doses | 14 | 21 | 10 | 16 | 20
  Grade 3 Muscle aches, Across doses | 0 | 1 | 1 | 0 | 2
  Related Muscle aches, Across doses | 13 | 17 | 9 | 13 | 16
  Any Shivering, Across doses | 4 | 5 | 3 | 3 | 7
  Grade 3 Shivering, Across doses | 0 | 1 | 0 | 0 | 1
  Related Shivering, Across doses | 4 | 2 | 2 | 0 | 4
  Any Sweating, Across doses | 2 | 5 | 5 | 3 | 7
  Grade 3 Sweating, Across doses | 0 | 0 | 1 | 0 | 2
  Related Sweating, Across doses | 2 | 4 | 3 | 2 | 5

6. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Laboratory Values
Description: Among analysed biochemical parameters were alanine aminotransferase [ALT], aspartate aminotransferase [AST], basophils [BAS], creatinine [CRE], eosinophils [EOS], hematocrit [HEM], hemoglobin [HgB], lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelets [PLA], red blood cells [RBC] and white blood cells [WBC].
Time Frame: At Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants
  ALT- Below | 0 | 0 | 0 | 0 | 0
  ALT- Above | 1 | 4 | 0 | 1 | 5
  AST- Below | 0 | 0 | 0 | 0 | 0
  AST- Above | 1 | 2 | 0 | 0 | 1
  BAS- Below | 0 | 0 | 0 | 0 | 0
  BAS- Above | 0 | 0 | 0 | 0 | 0
  CRE- Below | 1 | 6 | 6 | 7 | 8
  CRE- Above | 1 | 5 | 4 | 1 | 9
  EOS- Below | 3 | 2 | 8 | 4 | 13
  EOS- Above | 1 | 0 | 0 | 3 | 4
  HEM- Below | 0 | 0 | 2 | 2 | 1
  HEM- Above | 4 | 4 | 3 | 2 | 9
  HgB- Below | 1 | 0 | 2 | 3 | 1
  HgB- Above | 1 | 0 | 0 | 0 | 1
  LYM- Below | 1 | 0 | 0 | 2 | 2
  LYM- Above | 0 | 1 | 0 | 1 | 1
  MON- Below | 2 | 0 | 3 | 3 | 6
  MON- Above | 0 | 0 | 0 | 0 | 0
  NEU- Below | 0 | 0 | 0 | 0 | 1
  NEU- Above | 1 | 1 | 0 | 0 | 1
  PLA- Below | 0 | 0 | 1 | 0 | 4
  PLA- Above | 0 | 1 | 0 | 1 | 2
  RBC- Below | 0 | 1 | 2 | 0 | 0
  RBC- Above | 1 | 0 | 2 | 0 | 1
  WBC- Below | 1 | 0 | 0 | 0 | 3
  WBC- Above | 1 | 2 | 1 | 0 | 4

7. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Laboratory Values
Description: as for outcome 6
Time Frame: At Day 7
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects for whom safety data were available at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 59 | 60 | 60 | 59 | 120
Participants
  ALT- Below | 0 | 0 | 0 | 0 | 0
  ALT- Above | 1 | 3 | 1 | 1 | 2
  AST- Below | 0 | 0 | 0 | 0 | 0
  AST- Above | 1 | 2 | 1 | 0 | 1
  BAS- Below | 0 | 0 | 0 | 0 | 0
  BAS- Above | 0 | 0 | 0 | 0 | 0
  CRE- Below | 2 | 5 | 5 | 6 | 5
  CRE- Above | 2 | 5 | 3 | 0 | 8
  EOS- Below | 3 | 2 | 7 | 5 | 10
  EOS- Above | 0 | 0 | 2 | 2 | 3
  HEM- Below | 2 | 1 | 2 | 1 | 2
  HEM- Above | 1 | 2 | 1 | 1 | 6
  HgB- Below | 2 | 1 | 4 | 2 | 2
  HgB- Above | 0 | 0 | 0 | 0 | 0
  LYM- Below | 3 | 0 | 1 | 1 | 2
  LYM- Above | 0 | 1 | 0 | 1 | 2
  MON- Below | 2 | 0 | 3 | 7 | 6
  MON- Above | 0 | 0 | 0 | 0 | 1
  NEU- Below | 2 | 0 | 0 | 0 | 0
  NEU- Above | 0 | 0 | 1 | 0 | 3
  PLA- Below | 0 | 0 | 1 | 1 | 5
  PLA- Above | 0 | 1 | 0 | 1 | 3
  RBC- Below | 1 | 0 | 2 | 1 | 1
  RBC- Above | 0 | 0 | 1 | 0 | 0
  WBC- Below | 0 | 1 | 0 | 0 | 2
  WBC- Above | 0 | 1 | 0 | 1 | 3

8. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Laboratory Values
Description: as for outcome 6
Time Frame: At Day 21
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects for whom safety data were available at Day 21.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 119
Participants
  ALT- Below | 0 | 0 | 0 | 0 | 0
  ALT- Above | 2 | 4 | 1 | 3 | 3
  AST- Below | 0 | 0 | 0 | 0 | 0
  AST- Above | 1 | 3 | 0 | 0 | 3
  BAS- Below | 0 | 0 | 0 | 0 | 0
  BAS- Above | 0 | 0 | 0 | 0 | 0
  CRE- Below | 0 | 6 | 5 | 6 | 7
  CRE- Above | 4 | 4 | 3 | 1 | 9
  EOS- Below | 2 | 2 | 7 | 7 | 8
  EOS- Above | 1 | 0 | 1 | 2 | 4
  HEM- Below | 0 | 1 | 3 | 5 | 2
  HEM- Above | 0 | 2 | 2 | 2 | 4
  HgB- Below | 1 | 1 | 3 | 4 | 4
  HgB- Above | 0 | 0 | 0 | 0 | 2
  LYM- Below | 1 | 0 | 0 | 1 | 3
  LYM- Above | 0 | 1 | 1 | 0 | 1
  MON- Below | 4 | 5 | 3 | 4 | 10
  MON- Above | 0 | 0 | 1 | 0 | 0
  NEU- Below | 1 | 0 | 0 | 0 | 0
  NEU- Above | 0 | 1 | 1 | 0 | 2
  PLA- Below | 0 | 0 | 1 | 1 | 5
  PLA- Above | 0 | 1 | 0 | 1 | 3
  RBC- Below | 0 | 0 | 3 | 1 | 3
  RBC- Above | 0 | 1 | 1 | 0 | 0
  WBC- Below | 1 | 1 | 0 | 0 | 2
  WBC- Above | 1 | 2 | 1 | 0 | 2

9. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Laboratory Values
Description: as for outcome 6
Time Frame: At Day 28
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects for whom safety data were available at Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 118
Participants
  ALT- Below | 0 | 0 | 0 | 0 | 0
  ALT-Above | 1 | 2 | 1 | 0 | 3
  AST- Below | 0 | 0 | 0 | 0 | 0
  AST- Above | 1 | 1 | 1 | 0 | 2
  BAS- Below | 0 | 0 | 0 | 0 | 0
  BAS- Above | 0 | 0 | 0 | 0 | 0
  CRE- Below | 0 | 4 | 3 | 4 | 2
  CRE- Above | 2 | 2 | 3 | 2 | 8
  EOS- Below | 2 | 6 | 5 | 3 | 9
  EOS- Above | 2 | 1 | 1 | 2 | 2
  HEM- Below | 1 | 2 | 3 | 4 | 3
  HEM- Above | 2 | 0 | 1 | 0 | 2
  HgB- Below | 2 | 2 | 4 | 4 | 4
  HgB- Above | 1 | 0 | 0 | 0 | 1
  LYM- Below | 2 | 0 | 0 | 1 | 3
  LYM- Above | 2 | 1 | 0 | 0 | 0
  MON- Below | 3 | 2 | 5 | 3 | 8
  MON- Above | 0 | 1 | 0 | 0 | 0
  NEU- Below | 1 | 1 | 1 | 0 | 0
  NEU- Above | 0 | 2 | 1 | 0 | 0
  PLA- Below | 0 | 0 | 1 | 1 | 4
  PLA- Above | 0 | 1 | 0 | 3 | 3
  RBC- Below | 0 | 0 | 3 | 2 | 3
  RBC- Above | 1 | 0 | 1 | 0 | 0
  WBC- Below | 0 | 0 | 1 | 0 | 2
  WBC- Above | 1 | 2 | 1 | 3 | 1

10. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Laboratory Values
Description: as for outcome 6
Time Frame: At Day 42
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects for whom safety data were available at Day 42.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 118
Participants
  ALT- Below: number analyzed (Participants) | 58 | 60 | 60 | 60 | 118
  ALT- Below | 0 | 0 | 0 | 0 | 0
  ALT- Above: number analyzed (Participants) | 58 | 60 | 60 | 60 | 118
  ALT- Above | 1 | 4 | 1 | 0 | 6
  AST- Below | 0 | 0 | 0 | 0 | 0
  AST- Above | 1 | 1 | 1 | 0 | 2
  BAS- Below | 0 | 0 | 0 | 0 | 0
  BAS- Above | 0 | 0 | 0 | 0 | 0
  CRE- Below | 0 | 7 | 3 | 3 | 7
  CRE- Above | 3 | 4 | 5 | 3 | 8
  EOS- Below | 3 | 6 | 9 | 3 | 10
  EOS- Above | 1 | 0 | 1 | 2 | 3
  HEM- Below | 1 | 1 | 3 | 4 | 3
  HEM- Above | 1 | 1 | 3 | 1 | 2
  HgB- Below | 1 | 1 | 5 | 3 | 3
  HgB- Above | 0 | 0 | 0 | 0 | 1
  LYM- Below | 1 | 1 | 0 | 0 | 4
  LYM- Above | 0 | 0 | 0 | 1 | 0
  MON- Below | 2 | 10 | 5 | 8 | 18
  MON- Above | 1 | 0 | 0 | 0 | 0
  NEU- Below | 0 | 0 | 0 | 0 | 0
  NEU- Above | 1 | 0 | 1 | 1 | 3
  PLA- Below | 0 | 0 | 1 | 2 | 5
  PLA- Above | 0 | 1 | 0 | 2 | 3
  RBC- Below | 0 | 0 | 1 | 2 | 1
  RBC- Above | 1 | 0 | 2 | 0 | 0
  WBC- Below | 0 | 1 | 0 | 0 | 2
  WBC- Above | 2 | 1 | 1 | 1 | 2

11. Primary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 up to Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 2 | 10 | 7 | 3 | 16

12. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: Any pIMD was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 1 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 up to Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 17 | 18 | 21 | 17 | 35

14. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 0 | 3 | 1 | 1 | 2

15. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value for Vaccine-homologous (H7N1)
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 0, 21, 42 and Months 6 and 12
Population: The analysis was performed on the adapted According-to-Protocol cohort for immunogenicity, which included all evaluable subjects for which Days 0, 21, and 42 data were obtained from the ATP cohort for immunogenicity at Day 42; Months 6 and 12 data were obtained from the ATP cohorts for immunogenicity at Months 6 and 12 respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 57 | 55 | 53 | 114
Participants
  Flu A/mallard/NL/12/2000 (H7N1), Day 0: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 0 | 0 | 4 | 3 | 1 | 3
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 16 | 18 | 25 | 23 | 4
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 56 | 56 | 55 | 53 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 47 | 56 | 50 | 48 | 7
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 56 | 57 | 54 | 51 | 114
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 25 | 37 | 35 | 38 | 4
  Flu A/mallard/NL/12/2000 (H7N1), Month 12: number analyzed (Participants) | 51 | 55 | 51 | 46 | 106
  Flu A/mallard/NL/12/2000 (H7N1), Month 12 | 4 | 7 | 9 | 10 | 1

16. Secondary Outcome: Titers for Antibodies Against Flu A/Mallard/NL/12/2000 Strain of Influenza Disease Vaccine-homologous (H7N1)
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 0, 21, 42 and Months 6 and 12
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 57 | 55 | 53 | 114
Titers
  Flu A/mallard/NL/12/2000 (H7N1), Day 0: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 0 | 5.0 [5.0 to 5.0] | 5.6 [5.0 to 6.4] | 5.4 [4.9 to 5.8] | 5.1 [4.9 to 5.4] | 5.2 [5.0 to 5.5]
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 8.2 [6.5 to 10.2] | 8.9 [7.0 to 11.3] | 11.1 [8.6 to 14.5] | 10.6 [8.2 to 13.5] | 5.3 [5.0 to 5.6]
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 56 | 56 | 55 | 53 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 55.0 [36.7 to 82.5] | 104.8 [80.3 to 136.7] | 85.5 [58.0 to 126.1] | 97.0 [67.5 to 139.4] | 5.4 [5.1 to 5.8]
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 56 | 57 | 54 | 51 | 114
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 10.7 [8.4 to 13.7] | 16.1 [12.6 to 20.5] | 17.1 [12.9 to 22.6] | 17.5 [13.7 to 22.2] | 5.2 [5.0 to 5.5]
  Flu A/mallard/NL/12/2000 (H7N1), Month 12: number analyzed (Participants) | 51 | 55 | 51 | 46 | 106
  Flu A/mallard/NL/12/2000 (H7N1), Month 12 | 5.7 [5.0 to 6.4] | 5.9 [5.2 to 6.8] | 6.6 [5.6 to 7.9] | 7.2 [5.7 to 8.9] | 5.0 [5.0 to 5.1]

17. Secondary Outcome: Number of Seroprotected (SPR) Subjects Against HI Antibodies for Vaccine-homologous (H7N1)
Description: Seroprotection (SPR) was defined as the proportion of subjects with H7N1 reciprocal HI titers equal to or above (≥) 1:40 against the tested vaccine virus. The flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 0, 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 57 | 55 | 53 | 114
Participants
  Flu A/mallard/NL/12/2000 (H7N1), Day 0: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 0 | 0 | 1 | 0 | 0 | 1
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 7 | 6 | 9 | 8 | 1
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 56 | 56 | 55 | 53 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 39 | 49 | 43 | 47 | 1
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 56 | 57 | 54 | 51 | 114
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 10 | 17 | 17 | 14 | 0
  Flu A/mallard/NL/12/2000 (H7N1), Month 12: number analyzed (Participants) | 51 | 55 | 51 | 46 | 106
  Flu A/mallard/NL/12/2000 (H7N1), Month 12 | 2 | 1 | 1 | 3 | 0

18. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies for Vaccine-homologous (H7N1)
Description: SCR was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 55 | 55 | 52 | 113
Participants
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 7 | 4 | 9 | 8 | 0
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 39 | 45 | 42 | 46 | 0
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 56 | 55 | 54 | 50 | 113
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 10 | 15 | 15 | 14 | 0
  Flu A/mallard/NL/12/2000 (H7N1), Month 12: number analyzed (Participants) | 51 | 55 | 51 | 46 | 106
  Flu A/mallard/NL/12/2000 (H7N1), Month 12 | 2 | 1 | 1 | 3 | 0

19. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/Mallard/NL/12/2000 Strain of Influenza Disease Vaccine-homologous (H7N1)
Description: GMFR, also known as seroconversion factor (SCF), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus. The flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 56 | 55 | 55 | 52 | 113
Fold increase
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 1.6 [1.3 to 2.0] | 1.6 [1.3 to 1.9] | 2.1 [1.6 to 2.7] | 2.1 [1.6 to 2.6] | 1.0 [1.0 to 1.0]
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 56 | 55 | 55 | 52 | 112
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 11.0 [7.3 to 16.5] | 18.9 [14.0 to 25.4] | 16.0 [10.8 to 23.7] | 18.2 [12.6 to 26.3] | 1.0 [1.0 to 1.1]
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 56 | 55 | 54 | 50 | 113
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 2.1 [1.7 to 2.7] | 3.0 [2.3 to 3.8] | 3.2 [2.4 to 4.2] | 3.4 [2.7 to 4.4] | 1.0 [1.0 to 1.1]
  Flu A/mallard/NL/12/2000 (H7N1), Month 12: number analyzed (Participants) | 51 | 55 | 51 | 46 | 106
  Flu A/mallard/NL/12/2000 (H7N1), Month 12 | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.3] | 1.3 [1.1 to 1.5] | 1.4 [1.1 to 1.8] | 1.0 [0.9 to 1.0]

20. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value for Vaccine-heterologous (H7N9)
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/Shanghai/2/2013 (H7N9).
Time Frame: At Days 0, 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 28 | 29 | 25 | 30
Participants
  Flu A/Shanghai/2/2013 (H7N9), Day 0: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 0 | 0 | 1 | 1 | 2 | 1
  Flu A/Shanghai/2/2013 (H7N9), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 21 | 6 | 13 | 12 | 9 | 1
  Flu A/Shanghai/2/2013 (H7N9), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 42 | 24 | 27 | 24 | 24 | 1
  Flu A/Shanghai/2/2013 (H7N9), Month 6: number analyzed (Participants) | 28 | 28 | 28 | 23 | 29
  Flu A/Shanghai/2/2013 (H7N9), Month 6 | 10 | 19 | 18 | 14 | 0
  Flu A/Shanghai/2/2013 (H7N9), Month 12: number analyzed (Participants) | 24 | 28 | 26 | 20 | 23
  Flu A/Shanghai/2/2013 (H7N9), Month 12 | 2 | 11 | 11 | 4 | 1

21. Secondary Outcome: Titers for Antibodies Against Flu A/Shanghai/2/2013 Strain of Influenza Disease Vaccine-heterologous (H7N9)
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was Flu A/Shanghai/2/2013 (H7N9).
Time Frame: At Days 0, 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 28 | 29 | 25 | 30
Titers
  Flu A/Shanghai/2/2013 (H7N9), Day 0: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 0 | 5.0 [5.0 to 5.0] | 5.3 [4.7 to 6.1] | 5.2 [4.8 to 5.8] | 5.8 [4.7 to 7.1] | 5.2 [4.8 to 5.8]
  Flu A/Shanghai/2/2013 (H7N9), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 21 | 7.6 [5.4 to 10.7] | 12.5 [8.2 to 18.9] | 10.0 [7.1 to 13.9] | 10.9 [6.8 to 17.4] | 5.2 [4.8 to 5.8]
  Flu A/Shanghai/2/2013 (H7N9), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 42 | 64.3 [36.6 to 113.2] | 201.3 [142.6 to 284.1] | 96.4 [51.6 to 179.9] | 179.9 [103.1 to 314.0] | 5.2 [4.8 to 5.8]
  Flu A/Shanghai/2/2013 (H7N9), Month 6: number analyzed (Participants) | 28 | 28 | 28 | 23 | 29
  Flu A/Shanghai/2/2013 (H7N9), Month 6 | 8.6 [6.4 to 11.6] | 14.1 [10.4 to 19.1] | 14.7 [10.3 to 20.9] | 12.6 [8.9 to 17.7] | 5.0 [5.0 to 5.0]
  Flu A/Shanghai/2/2013 (H7N9), Month 12: number analyzed (Participants) | 24 | 28 | 26 | 20 | 23
  Flu A/Shanghai/2/2013 (H7N9), Month 12 | 5.6 [4.8 to 6.6] | 8.4 [6.3 to 11.1] | 9.0 [6.5 to 12.3] | 7.0 [4.7 to 10.4] | 5.4 [4.6 to 6.2]

22. Secondary Outcome: Number of Seroprotected (SPR) Subjects Against HI Antibodies for Vaccine-heterologous (H7N9)
Description: Seroprotection (SPR) was defined as the proportion of subjects with H7N9 reciprocal HI titers equal to or above (≥) 1:40 against the tested vaccine virus. The flu strain assessed was Flu A/Shanghai/2/2013 (H7N9).
Time Frame: At Days 0, 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 28 | 29 | 25 | 30
Participants
  Flu A/Shanghai/2/2013 (H7N9), Day 0: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 0 | 0 | 0 | 0 | 1 | 0
  Flu A/Shanghai/2/2013 (H7N9), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 21 | 2 | 9 | 4 | 6 | 0
  Flu A/Shanghai/2/2013 (H7N9), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 42 | 22 | 26 | 23 | 23 | 0
  Flu A/Shanghai/2/2013 (H7N9), Month 6: number analyzed (Participants) | 28 | 28 | 28 | 23 | 29
  Flu A/Shanghai/2/2013 (H7N9), Month 6 | 2 | 5 | 6 | 3 | 0
  Flu A/Shanghai/2/2013 (H7N9), Month 12: number analyzed (Participants) | 24 | 28 | 26 | 20 | 23
  Flu A/Shanghai/2/2013 (H7N9), Month 12 | 0 | 3 | 2 | 1 | 0

23. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies for Vaccine-heterologous (H7N9)
Description: SCR was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strain assessed was Flu A/Shanghai/2/2013 (H7N9).
Time Frame: At Days 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 27 | 28 | 29 | 24 | 30
Participants
  Flu A/Shanghai/2/2013 (H7N9), Day 21: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 21 | 2 | 8 | 3 | 4 | 0
  Flu A/Shanghai/2/2013 (H7N9), Day 42: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 42 | 22 | 26 | 23 | 22 | 0
  Flu A/Shanghai/2/2013 (H7N9), Month 6: number analyzed (Participants) | 27 | 28 | 28 | 22 | 29
  Flu A/Shanghai/2/2013 (H7N9), Month 6 | 2 | 5 | 6 | 2 | 0
  Flu A/Shanghai/2/2013 (H7N9), Month 12: number analyzed (Participants) | 24 | 28 | 26 | 20 | 23
  Flu A/Shanghai/2/2013 (H7N9), Month 12 | 0 | 3 | 2 | 1 | 0

24. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/Shanghai/2/2013 Strain of Influenza Disease Vaccine-heterologous (H7N9)
Description: GMFR, also known as seroconversion factor (SCF), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus. The flu strain assessed was Flu A/Shanghai/2/2013 (H7N9).
Time Frame: At Days 21 and 42 and at Months 6 and 12
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 27 | 28 | 29 | 24 | 30
Fold increase
  Flu A/Shanghai/2/2013 (H7N9), Day 21: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 21 | 1.5 [1.1 to 2.2] | 2.3 [1.6 to 3.5] | 1.9 [1.4 to 2.6] | 1.7 [1.1 to 2.5] | 1.0 [1.0 to 1.0]
  Flu A/Shanghai/2/2013 (H7N9), Day 42: number analyzed (Participants) | 27 | 27 | 29 | 24 | 30
  Flu A/Shanghai/2/2013 (H7N9), Day 42 | 14.1 [8.1 to 24.6] | 37.7 [25.8 to 54.9] | 18.4 [9.8 to 34.4] | 28.7 [15.6 to 52.7] | 1.0 [1.0 to 1.0]
  Flu A/Shanghai/2/2013 (H7N9), Month 6: number analyzed (Participants) | 27 | 28 | 28 | 22 | 29
  Flu A/Shanghai/2/2013 (H7N9), Month 6 | 1.8 [1.3 to 2.4] | 2.6 [1.9 to 3.6] | 2.8 [2.0 to 4.0] | 2.0 [1.3 to 3.2] | 1.0 [0.9 to 1.1]
  Flu A/Shanghai/2/2013 (H7N9), Month 12: number analyzed (Participants) | 24 | 28 | 26 | 20 | 23
  Flu A/Shanghai/2/2013 (H7N9), Month 12 | 1.1 [1.0 to 1.3] | 1.6 [1.2 to 2.1] | 1.7 [1.2 to 2.3] | 1.2 [0.7 to 1.9] | 1.0 [0.8 to 1.2]

25. Secondary Outcome: Number of Subjects With HI Neutralizing Antibody Concentrations Above the Cut-off Value for Vaccine-homologous (H7N1)
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:28 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 0, 21 and 42 and Month 6
Population: The analysis was performed on the adapted According-to-Protocol cohort for immunogenicity, which included all evaluable subjects for which Days 0, 21, and 42 data were obtained from the ATP cohort for immunogenicity at Day 42; Month 6 data was obtained from the ATP cohort for immunogenicity at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 29 | 29 | 25 | 30
Participants
  Flu A/mallard/NL/12/2000 (H7N1), Day 0: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 0 | 2 | 7 | 3 | 2 | 3
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 9 | 13 | 9 | 12 | 2
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 26 | 27 | 24 | 24 | 2
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 28 | 29 | 28 | 23 | 29
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 22 | 27 | 23 | 20 | 3

26. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Mallard/NL/12/2000 Strain of Influenza Disease Vaccine-homologous (H7N1)
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/mallard/NL/12/2000. The reference seropositivity cut-off value was ≥ 1:28.
Time Frame: At Days 0, 21 and 42 and at Month 6
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 29 | 29 | 25 | 30
Titers
  Flu A/mallard/NL/12/2000 (H7N1), Day 0: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 0 | 14.7 [13.7 to 15.8] | 16.8 [14.8 to 18.9] | 15.0 [13.9 to 16.3] | 14.8 [13.7 to 16.0] | 15.0 [13.9 to 16.2]
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 17.5 [15.4 to 19.9] | 21.2 [17.5 to 25.6] | 18.2 [15.5 to 21.5] | 21.9 [17.6 to 27.2] | 14.7 [13.7 to 15.7]
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 46.2 [34.2 to 62.5] | 71.4 [56.8 to 89.7] | 51.3 [38.1 to 69.1] | 74.7 [54.2 to 102.9] | 14.7 [13.7 to 15.7]
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 28 | 29 | 28 | 23 | 29
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 26.7 [22.7 to 31.5] | 38.5 [32.1 to 46.3] | 33.5 [27.0 to 41.7] | 39.4 [31.6 to 49.3] | 15.0 [13.9 to 16.3]

27. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Against the Flu A/Mallard/NL/12/2000 (H7N1) Virus Strain
Description: Vaccine response was defined as: For initially seronegative subjects antibody titer ≥ 1:56 at post-vaccination]; For initially seropositive subjects antibody titer at post-vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/mallard/NL/12/2000 (H7N1).
Time Frame: At Days 21 and 42 and at Month 6
Population: The analysis was performed on the adapted According-to-Protocol cohort for immunogenicity, which included all evaluable subjects for which Days 21 and 42 data were obtained from the ATP cohort for immunogenicity at Day 42; Month 6 data was obtained from the ATP cohort for immunogenicity at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 29 | 29 | 25 | 30
Participants
  Flu A/mallard/NL/12/2000 (H7N1), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 21 | 0 | 0 | 1 | 3 | 0
  Flu A/mallard/NL/12/2000 (H7N1), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/mallard/NL/12/2000 (H7N1), Day 42 | 13 | 22 | 17 | 19 | 0
  Flu A/mallard/NL/12/2000 (H7N1), Month 6: number analyzed (Participants) | 28 | 29 | 28 | 23 | 29
  Flu A/mallard/NL/12/2000 (H7N1), Month 6 | 4 | 9 | 10 | 13 | 0

28. Secondary Outcome: Number of Subjects With HI Neutralizing Antibody Concentrations Above the Cut-off Value for Vaccine-heterologous (H7N9)
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:28 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/Anhui/1/2013 (H7N9).
Time Frame: At Days 0, 21 and 42 and at Month 6
Population: The analysis was performed on the adapted According-to-Protocol cohort for immunogenicity, which included all evaluable subjects for which Days 0, 21 and 42 data were obtained from the ATP cohort for immunogenicity at Day 42; Month 6 data was obtained from the ATP cohort for immunogenicity at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 29 | 29 | 25 | 30
Participants
  Flu A/Anhui/1/2013 (H7N9), Day 0: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 0 | 0 | 1 | 0 | 2 | 0
  Flu A/Anhui/1/2013 (H7N9), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 21 | 3 | 12 | 7 | 12 | 0
  Flu A/Anhui/1/2013 (H7N9), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 42 | 25 | 27 | 23 | 24 | 0
  Flu A/Anhui/1/2013 (H7N9), Month 6: number analyzed (Participants) | 28 | 29 | 28 | 23 | 29
  Flu A/Anhui/1/2013 (H7N9), Month 6 | 16 | 23 | 22 | 20 | 1

29. Secondary Outcome: Titers for Antibodies Against Flu A/Anhui/1/2013 Strain of Influenza Disease Vaccine-homologous (H7N9)
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/Anhui/1/2013. The reference seropositivity cut-off value was ≥ 1:28.
Time Frame: At Days 0, 21 and 42 and at Month 6
Population: as for outcome 25
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 29 | 29 | 25 | 30
Titers
  Flu A/Anhui/1/2013 (H7N9), Day 0: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 0 | 14.0 [14.0 to 14.0] | 14.4 [13.6 to 15.1] | 14.0 [14.0 to 14.0] | 14.8 [13.7 to 16.0] | 14.0 [14.0 to 14.0]
  Flu A/Anhui/1/2013 (H7N9), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 21 | 15.1 [13.9 to 16.4] | 20.1 [16.8 to 24.0] | 16.5 [14.8 to 18.6] | 21.3 [17.3 to 26.1] | 14.0 [14.0 to 14.0]
  Flu A/Anhui/1/2013 (H7N9), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 42 | 44.0 [32.4 to 59.7] | 79.1 [60.5 to 103.3] | 53.8 [37.8 to 76.6] | 85.6 [60.9 to 120.5] | 14.0 [14.0 to 14.0]
  Flu A/Anhui/1/2013 (H7N9), Month 6: number analyzed (Participants) | 28 | 29 | 28 | 23 | 30
  Flu A/Anhui/1/2013 (H7N9), Month 6 | 24.8 [19.6 to 31.4] | 34.2 [27.3 to 42.8] | 36.1 [27.6 to 47.3] | 35.9 [28.9 to 44.7] | 14.3 [13.7 to 15.1]

30. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Against the Flu A/Anhui/1/2013 (H7N9) Virus Strain
Description: Vaccine response was defined as: For initially seronegative subjects antibody titer ≥ 1:56 at post-vaccination]; For initially seropositive subjects antibody titer at post-vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/Anhui/1/2013 (H7N9).
Time Frame: At Days 21 and 42 and at Month 6
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 28 | 29 | 29 | 25 | 30
Participants
  Flu A/Anhui/1/2013 (H7N9), Day 21: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 21 | 0 | 2 | 0 | 3 | 0
  Flu A/Anhui/1/2013 (H7N9), Day 42: number analyzed (Participants) | 28 | 27 | 29 | 25 | 30
  Flu A/Anhui/1/2013 (H7N9), Day 42 | 13 | 23 | 18 | 18 | 0
  Flu A/Anhui/1/2013 (H7N9), Month 6: number analyzed (Participants) | 28 | 29 | 28 | 23 | 29
  Flu A/Anhui/1/2013 (H7N9), Month 6 | 6 | 12 | 13 | 11 | 0

31. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination. Analysis of intensity and relationship to vaccination of MAEs was not performed.
Time Frame: From Day 42 up to Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 23 | 24 | 26 | 21 | 43

32. Secondary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: An pIMD was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 42 up to Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 0 | 0 | 0 | 1 | 0

33. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 13
Time Frame: During the 21-day (From Day 0 to Day 20) post-vaccination period after each dose
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 18 | 17 | 22 | 17 | 38

34. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 14
Time Frame: During the entire study period (From Day 0 up to Month 12)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 120
Participants | 3 | 10 | 7 | 7 | 13

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 21-day (Days 0-20) post-vaccination period after each dose; SAEs: during the entire study period (from Day 0 up to Month 12).
Arm/Group | GSK2789869A F1 Group | GSK2789869A F2 Group | GSK2789869A F3 Group | GSK2789869A F4 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/60 | 2/60 | 0/60 | 0/120
Serious Adverse Events (participants affected / at risk) | 3/60 | 10/60 | 7/60 | 7/60 | 13/120
Other Adverse Events (participants affected / at risk) | 46/60 | 48/60 | 30/60 | 44/60 | 47/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2789869A F1 Group (N=60) | GSK2789869A F2 Group (N=60) | GSK2789869A F3 Group (N=60) | GSK2789869A F4 Group (N=60) | Placebo Group (N=120)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2789869A F1 Group (N=60) | GSK2789869A F2 Group (N=60) | GSK2789869A F3 Group (N=60) | GSK2789869A F4 Group (N=60) | Placebo Group (N=120)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Pain (General disorders) | 38 (54) | 39 (58) | 25 (33) | 38 (54) | 9 (11)
Redness (General disorders) | 1 (1) | 4 (4) | 1 (2) | 4 (4) | 1 (1)
Swelling (General disorders) | 2 (2) | 2 (3) | 4 (5) | 2 (2) | 0 (0)
Fatigue (General disorders) | 11 (14) | 19 (25) | 13 (17) | 11 (15) | 28 (35)
Gastrointestinal (General disorders) | 11 (12) | 11 (13) | 8 (11) | 9 (9) | 16 (18)
Headache (General disorders) | 13 (18) | 17 (26) | 13 (20) | 11 (15) | 24 (31)
Joint pain (General disorders) | 12 (13) | 13 (15) | 8 (10) | 9 (13) | 17 (25)
Muscle aches (General disorders) | 14 (20) | 21 (25) | 10 (13) | 16 (22) | 21 (30)
Shivering (Chills) (General disorders) | 4 (6) | 5 (6) | 4 (5) | 3 (3) | 7 (8)
Sweating (General disorders) | 2 (3) | 5 (6) | 5 (7) | 3 (5) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.